CLINICAL TRIAL: NCT06236217
Title: Prediction of Spinal Anesthesia-Induced Hypotension in Cesarian Section: Carotid Artery-Corrected Flow Time Versus Cardiometry: Randomized Controlled Trial
Brief Title: Prediction of Spinal Anesthesia-Induced Hypotension in Cesarian Section: Carotid Artery-Corrected Flow Time Versus Cardiometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Shehab, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34801/07/21
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Spinal Anesthesia; Hypotension; Cesarian Section; Carotid Artery; Corrected Flow Time; Cardiometry
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Patients received standard of care with no intervention before spinal anesthesia.
- Carotid Ultrasound group (Experimental): The carotid artery corrected flow time (FTc) was used in patients to optimize the volume status before performing spinal anesthesia.
  Interventions: Other: Carotid Ultrasound
- Electrical cardiometry group (Experimental): Stroke volume variation (SVV) measured by electrical cardiometry (EC) was used to optimize the volume status before performing spinal anesthesia.
  Interventions: Other: Electrical cardiometry

INTERVENTIONS:
Other: Carotid Ultrasound — The carotid artery corrected flow time (FTc) was used in patients to optimize the volume status before performing spinal anesthesia.
  Arms: Carotid Ultrasound group
Other: Electrical cardiometry — Stroke volume variation (SVV) measured by electrical cardiometry (EC) was used to optimize the volume status before performing spinal anesthesia.
  Arms: Electrical cardiometry group

SUMMARY:
This research aimed to evaluate and compare the role of carotid corrected flow time (FTc) and electrical cardiometry (EC) in the prediction and prevention of post-spinal hypotension in elective cesarian section.

DETAILED DESCRIPTION:
Spinal anesthesia is the procedure of choice for elective cesarean section (CS) because it avoids the most common side effects related to general anesthesia, such as the risk of aspiration, airway problems and the negative effects of intravenous anesthetic drugs on the fetus.

Accurate prediction of post-spinal hypotension could enhance clinical decision-making, optimize management, and facilitate early intervention. More than thirty predictors were used in the prediction of post-spinal hypotension including demographic data, hemodynamic variables, postural stress testing, peripheral perfusion indices, volume and fluid responsiveness indices, and genetic polymorphism.

The baseline parameters obtained via the bioreactance-based system may serve as a predictor of post-spinal anesthesia hypotension in parturient.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* American Society of Anesthesiologists (ASA) physical status II.
* Gestational age (GA) ≥ 36 weeks.
* Women planned elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* Patient refusal to participate in the study.
* Gestational age of < 36 or ≥40 weeks of pregnancy.
* Pregnancy-induced hypertension.
* Diabetes.
* Cardiovascular diseases, arrhythmia.
* Antepartum hemorrhage.
* Body Mass Index (BMI) above 36 kg/m2.
* Clinical fetal complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women elective cesarean section
Enrollment: 300 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence of post-spinal hypotension | Intraoperatively
  Incidence of spinal anesthesia-induced hypotension was measured. Post spinal hypotension is defined as a drop in the SBP to less than 80mmHg, or less than 75% of the pre-anesthetic value. Hypotension was treated by IV vasopressor boluses (Ephedrine 5 mg).

SECONDARY OUTCOMES:
The amount of intravenous fluids | Intraoperatively
  The amount of intravenous fluids was assessed.
The amount of vasopressor | Intraoperatively
  The amount of vasopressor was assessed. Post spinal hypotension is defined as a drop in the SBP to less than 80mmHg, or less than 75% of the pre-anesthetic value. Hypotension was treated by IV vasopressor boluses (Ephedrine 5 mg).
Umbilical cord PH | Immediately after fetal delivery
  Umbilical cord PH was measured with fetal delivery.
Neonatal APGAR score | 5 minutes after fetal delivery
  Neonatal APGAR score is a score between 7-10 is normal; a score between 4-6 needs proper reevaluation as the infant does require monitoring for 5 minutes. It was measured at 1, 5 minutes.
Complications | Intraoperatively
  Complications such as bradycardia, pruritis and urine retention were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.